CLINICAL TRIAL: NCT01494324
Title: Examinations of Tissue From Ablated Malignant Liver Metastases as Predictors of Outcome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 09-122
Record Dates: First submitted 2011-12-13; First posted 2011-12-19 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Liver Cancer
Keywords: Liver; Thermal Ablation; Dynamic CT; 09-122
MeSH Terms: conditions — Liver Neoplasms | interventions — Long-Term Potentiation

ARMS (1):
- CT guided percutaneous ablation (Experimental): The selected patients will undergo CT guided percutaneous ablation. The use of multi-tined electrode is encouraged, unless tumor location requires the use of an internally cooled needle electrode to eliminate injury to an adjacent vital structure or the operator prefers to use an internally cooled electrode for a specific reason.
  Interventions: Other: CT guided percutaneous ablation

INTERVENTIONS:
Other: CT guided percutaneous ablation — Depending on tumor size and location, we will direct a core biopsy needle in the ablated tumor using post-ablation dynamic Liver CT guidance, preferably including liver triphasic examination. The obtained tissue will be detached, collected and submitted to our molecular cytology laboratory. All specimens will be submitted fresh to our molecular cytology laboratory for immediate analysis in order to classify them as viable tumor (V) or apoptotic cells/coagulation necrosis (CN). CT will be performed within 24 hours of the ablation to demonstrate the ablation defect, representing the area of coagulation necrosis. This CT will be used for targeting the ablated tumor for biopsy. All patients will undergo CT again, approximately within 4-8 weeks (+/- 2 weeks) of percutaneous ablation to evaluate for CN in the target tumor or any sign of residual tissue enhancement, representing incomplete treatment.
  Other Names: Follow-up will continue at approximate 2-4 months intervals (+/- 2 weeks) with CT, to evaluate for local tumor progression (LTP) for the following 3 years.

SUMMARY:
The purpose of this study is to see if the investigators can do some tests on tissue from the area of the ablation. The investigators want to know if a test can help predict whether the ablation worked.

The treated tumor is normally evaluated with CT. The CT shows signs of treated tumor(s) in the area treated by ablation. However, cancer cells may begin to grow in or near the treated area. The CT scan cannot tell us if the cells are new cancer cells or if they are healthy liver cells that just look different because of the ablation. The test the investigators will study should be able to tell us the difference.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed with secondary hepatic malignancy;
* Patients with confined liver disease or stable limited extrahepatic disease;
* Lesions of 5cm or less in maximum diameter;
* Patients who are not surgical candidates or refuse to undergo surgery and choose any percutaneous ablation as an alternative treatment option.
* INR<1.5 *for patients on Coumadin general clinical guidelines for IR ablation will be followed.
* Platelet count > or = to 50,000

Exclusion Criteria:

* Patients < 18
* Less than 5 mm distance of the tumor margin from a major vessel >7mm in diameter)**
* Less than 5 mm distance to a structure (GI or biliary tract), that cannot be protected from**
* the ablation injury with technical modifications such as hydro or air dissection.
* INR > 1.5 that cannot be corrected with fresh frozen Plasma*
* Platelet count of <50,000 that cannot be corrected with transfusion.
* Patient with more than 3 tumors treated with any percutaneous ablation
* Patients with more than 5 sites of extrahepatic disease (including nodes and pulmonary nodules)

  * for patients on Coumadin general clinical guidelines for IR ablation will be followed **This will not be considered an exclusion criteria when IRE or Microwave is used.

    * This will not be considered exclusion when IRE is used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-10-27 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Tumor response | 3 years
  will be measured according to EASL and RECIST. In the case of differences between these criteria, the EASL criteria will be used for clinical judgment and decisions.Tumor response will be determined at the discretion of the Principal Investigator in the case of overlapping ablation zones or lesions seen only in PET.

SECONDARY OUTCOMES:
Duration of treatment response | 3 years
  will be measured as the time from the date of first objective response until the first measurement of progression as determined by the central readers using the EASL criteria. Dynamic Liver CT scans, preferably including the liver triphasic examination will be conducted at each follow-up visit until progression.

CONTACTS AND LOCATIONS:
Overall Officials: Constantinos Sofocleous, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT01494324/ICF_000.pdf